CLINICAL TRIAL: NCT00820833
Title: Effect of Protein Levels and Caloric Density on the Growth of Formula Fed Infants From Overweight or Obese Mothers
Brief Title: Effect of Formula on Growth of Infants From Overweight or Obese Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 05.29.INF
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2014-12

CONDITIONS: Infant Nutrition
Keywords: infant formula; obesity; growth
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Standard infant formula
  Interventions: Other: standard infant formula
- 2 (Experimental): Test formula
  Interventions: Other: Test formula
- 3 (No Intervention): Breastfeeding reference group

INTERVENTIONS:
Other: standard infant formula — standard infant formula given from 3 to 12 months of age, as per standard requirement
  Arms: 1
Other: Test formula — Test formula with different protein and calorie content than standard formula, given from 3 to 12 months of age. As per standard requirement.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether infants, from overweight or obese mothers, fed a formula with proteins and calories different than a standard infant formula have a different growth

ELIGIBILITY:
Inclusion Criteria:

* healthy newborn infant
* birth weight between 2500g and 4800g
* singleton birth
* mother's BMI before pregnancy was between 26 and 25
* for the breastfeeding group: mother has elected to exclusively breastfeed her baby from birth to at least 6 months of age
* for the formula groups: mother has elected to exclusively formula feed her baby from 3 to 6 months of age
* having obtained signed informed consent of legal representative

Exclusion Criteria:

* body weight smaller than 5th percentile for that gestational age
* newborn whose mother has diabetes
* newborn whose mother has a drug dependence during pregnancy
* newborn currently participating in another trial

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2007-10; Primary Completion 2010-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
mean weight gain | 3 months

SECONDARY OUTCOMES:
blood test assessments; body composition, bone density | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Inostroza, PhD, Principal Investigator — Universidad de La Frontera
Locations (1):
- Departamento de Medicina Interna, University de la Frontera, Temuco, Chile

REFERENCES:
- [Derived] Inostroza J, Haschke F, Steenhout P, Grathwohl D, Nelson SE, Ziegler EE. Low-protein formula slows weight gain in infants of overweight mothers. J Pediatr Gastroenterol Nutr. 2014 Jul;59(1):70-7. doi: 10.1097/MPG.0000000000000349. PMID 24637965